CLINICAL TRIAL: NCT06675630
Title: Investigating Food Intake Across the Adult Life Course and Relevant Communication Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Principal Investigator, Stella Lignou, Associate Professor in Sensory and Consumer Science, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 26/2024
Record Dates: First submitted 2024-09-23; First posted 2024-11-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Individual Differences; Food Intake; Behaviour Change
Keywords: Lifecourse; Education; Fibre
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Healthy eating advice
  Interventions: Behavioral: Control
- Intervention (Experimental): Targeted fibre-related education
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Consumers will receive monthly targeted educational materials on fibre
  Arms: Intervention
Behavioral: Control — Consumers will receive educational materials on healthy eating at two timepoints
  Arms: Control

SUMMARY:
This project will investigate the effects of different delivery strategies (e.g., personalised dietary advice vs generalised population healthy eating guidance) and individual consumption differences (e.g., eating styles/speeds and food types/preferences) on dietary fibre intake across the adult life-course over a 6-month period.

DETAILED DESCRIPTION:
1. does dietary fibre-related knowledge and intake vary across the adult life-course?
2. what are the common barriers to dietary fibre consumption and how this modulates with increasing age?
3. what is the role of individual consumption differences on subsequent dietary fibre consumption?
4. can targeted dietary advice compared with general population healthy eating guidance delivered by the eNutri app promote dietary fibre intake?

ELIGIBILITY:
Inclusion Criteria

-adults aged 18 years and above

Exclusion Criteria

* health conditions impacting fibre intake (e.g., IBD, IBS, colorectal cancer, Crohns disease, ulcerative colitis, diverticulitis)
* pregnant or breastfeeding
* food allergies/intolerances
* following a weight-loss diet
* no digital device
* living outside of the UK
* cognition impairments (such as dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Food intake | One, three and six months (1-hr)
  Food intake will be measured via the eNutri app

SECONDARY OUTCOMES:
Food Consumption Differences | Visit one (1-hr)
  A series of validated questionnaires will measure the role of food-related consumption differences (e.g., foodie index, eating behaviour/rate, food preferences, mouth behaviour, food neophobia, knowledge, barriers, etc.) on subsequent food intake
Impact of Education | All visits (6-months)
  Education will vary depending on group allocation: (1) targeted fibre education will be circulated monthly; and (2) healthy eating advice will be shared twice during the study duration. Consumers will provide feedback on all materials at the end of the study
Fiberscreen tool | month 3 and 4
  Rate frequency of consumption of ten dietary fibre-rich food categories and estimate portion size

CONTACTS AND LOCATIONS:
Overall Officials: Stella Lignou (PI), Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Science, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Norton V, Lignou S, Methven L. Influence of Age and Individual Differences on Mouthfeel Perception of Whey Protein-Fortified Products: A Review. Foods. 2021 Feb 16;10(2):433. doi: 10.3390/foods10020433. PMID 33669435
- [Background] Zenun Franco R, Fallaize R, Lovegrove JA, Hwang F. Online dietary intake assessment using a graphical food frequency app (eNutri): Usability metrics from the EatWellUK study. PLoS One. 2018 Aug 10;13(8):e0202006. doi: 10.1371/journal.pone.0202006. eCollection 2018. PMID 30096211
- [Background] Norton V, Lovegrove JA, Tindall M, Garcia JR, Lignou S. Fibre4life: Investigating older adults dietary fibre preferences and the role of targeted educational materials on modulating future dietary fibre intake. Appetite. 2024 Jan 1;192:107109. doi: 10.1016/j.appet.2023.107109. Epub 2023 Oct 31. PMID 37914038
- [Background] Zenun Franco R, Fallaize R, Weech M, Hwang F, Lovegrove JA. Effectiveness of Web-Based Personalized Nutrition Advice for Adults Using the eNutri Web App: Evidence From the EatWellUK Randomized Controlled Trial. J Med Internet Res. 2022 Apr 25;24(4):e29088. doi: 10.2196/29088. PMID 35468093